CLINICAL TRIAL: NCT02330549
Title: ORION - Effect of CCR2 and CCR5 Antagonism by Cenicriviroc on Peripheral and Adipose Tissue Insulin Sensitivity in Adult Obese Subjects With Prediabetes or Type 2 Diabetes Mellitus and Suspected Non-Alcoholic Fatty Liver Disease (NAFLD)
Brief Title: ORION: Effects of Cenicriviroc on Insulin Sensitivity in Subjects With Prediabetes or Type 2 Diabetes Mellitus (T2DM) and Suspected NAFLD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tobira Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 652-2-204
Record Dates: First submitted 2014-12-22; First posted 2015-01-05 (Estimated); Results first posted 2019-10-11 (Actual); Last update posted 2019-10-11 (Actual); Status verified 2019-09

CONDITIONS: Prediabetic State; Non-alcoholic Fatty Liver Disease; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Prediabetic State; Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2 | interventions — cenicriviroc

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cenicriviroc 150 mg (Experimental): Cenicriviroc (CVC) 150 mg, administered orally once daily and taken every morning with food for up to 24 weeks.
  Interventions: Drug: Cenicriviroc 150 mg
- Placebo (Placebo Comparator): Placebo-matching CVC, administered orally once daily and taken every morning with food for up to 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cenicriviroc 150 mg — Cenicriviroc (CVC) 150 mg, administered orally once daily and taken every morning with food.
  Arms: Cenicriviroc 150 mg
Drug: Placebo — Placebo-matching CVC administered orally once daily and taken every morning with food.
  Arms: Placebo

SUMMARY:
A Phase 2a, randomized, double-blind, placebo-controlled, multi-center study of cenicriviroc (CVC) to be conducted in approximately 50 adult obese subjects [body mass index (BMI) ≥ 30 kg/m^2] with prediabetes or type 2 diabetes mellitus and suspected NALFD.

DETAILED DESCRIPTION:
Approximately 50 adult obese subjects (BMI ≥ 30 kg/m2) with prediabetes or type 2 diabetes mellitus and suspected NALFD will be randomized into the study.

Eligible subjects will receive either CVC (n=25) or matching placebo (n=25), once daily (QD) for 24 weeks, followed by a safety follow-up visit 4 weeks after last intake of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female subjects aged between 18-75 years
* Obesity as defined by BMI ≥ 30 kg/m2
* Evidence of prediabetes or type 2 diabetes mellitus based on Screening laboratory values with at least one of the following criteria:
* Fasting plasma glucose (FPG) of 100 - 270 mg/dL (5.6 - 15.0 mmol/L)
* Hemoglobin A1c (HbA1c) of 5.7 - 10.0%
* Participants receiving metformin alone or in combination with a sulfonylurea (glimepiride, glipizide, glyburide, or gliclazide) must be on stable therapy for at least 90 days prior to Screening.
* Suspected diagnosis of NAFLD warranting confirmation by liver biopsy
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 5 upper limit normal (ULN)
* Ability to understand and sign a written informed consent form
* Females of child-bearing potential and males participating in the study must agree to use at least 2 approved barrier methods of contraception throughout the duration of the study and for 3 months after stopping study drug. Females who are postmenopausal must have documentation of cessation of menses for ≥ 12 months and serum follicle stimulating hormone (FSH) ≥ 30 mU/mL
* Participants receiving allowed concomitant medications need to be on stable therapy for 28 days prior to Baseline.

Exclusion Criteria:

* Use of oral antihyperglycemic agents (OHAs) other than metformin or sulfonylureas, including but not limited to thiazolidinediones, DPP-4 inhibitors, SGLT2 inhibitors, GLP-1 receptor agonists, meglitinides, α-glucosidase inhibitors, colesevelam, bromocriptine, pramlintide or basal insulin within 90 days prior to Screening or anticipated use during the trial
* Type 1 diabetes
* Hepatitis B Surface Antigen (HBsAg) positive
* Human Immunodeficiency Virus-1 (HIV-1) or Human Immunodeficiency Virsu-2 (HIV-2) infection
* Hepatitis C Virus Antibody (HCVAb) positive
* Prior or planned liver transplantation
* Other known causes of chronic liver disease, including alcoholic liver disease
* History of cirrhosis and/or hepatic decompensation including ascites, encephalopathy or variceal bleeding
* Alcohol consumption greater than 14 units/week
* Weight reduction through bariatric surgery or planned bariatric surgery during the conduct of the study (including gastric banding)
* Any Grade ≥ 3 laboratory abnormality as defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Toxicity Grading Scale, except subjects with Grade ≥ 3 dyslipidemia with triglyceride or cholesterol elevations unless clinical assessment foresees an immediate health risk to the subject
* Serum albumin < 3.5 g/dL
* Serum creatinine levels ≥ 1.5 mg/dL for males or ≥ 1.4 mg/dL for females if participant is receiving metformin
* Estimated glomerular filtration rate (eGFR) < 50 mL/min/1.73 m2 according to the Modification of Diet in Renal Disease (MDRD) equation
* Platelet count < 100,000/mm3
* Hemoglobin < 12 g/dL for males or < 11 g/dL for females
* Females who are pregnant or breastfeeding
* Receiving ongoing therapy with any disallowed medication at Screening
* Allergy to the study drug or its components
* Any other clinically significant disorders or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing and protocol requirements.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-07-17 (Actual); Primary Completion 2016-08-11 (Actual); Study Completion 2016-09-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Lefebvre, MD, Study Director — Allergan
Locations (3):
- United States (2):
  - San Antonio Military Medical Center, Fort Sam Houston, Texas
  - Gastroenterology Consultants of San Antonio Digestive Research Center, San Antonio, Texas
- Fundacion de Investigacion, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cenicriviroc 150 mg | Placebo
Started | 20 | 25
Completed | 16 | 24
Not Completed | 4 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Subject withdrew consent | 2 | 1
Not completed — Failure to meet randomization criteria | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cenicriviroc 150 mg | Placebo | Total
Number analyzed (Participants) | 20 | 25 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (9.67) | 51.0 (8.98) | 52.2 (9.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 12 | 21
  Male | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Matsuda Index
Description: Change in peripheral insulin sensitivity was measured by the Matsuda Index. Fasting plasma glucose (FPG) and fasting plasma insulin (FPI) concentrations measured during the oral glucose tolerance test (OGTT) were used to calculate the Matsuda Index. Matsuda Index=10,000/square root [FPG mg/dL x FPI μIU/mL) x (mean glucose mg/dL x mean insulin μIU/mL during OGTT)]. A Matsuda index of <2.5 indicates whole body insulin resistance. A lower Matsuda Index indicates the worst disease state. An increase in the Matsuda Index indicates an improvement in insulin sensitivity (best). A positive change from Baseline indicates improvement and a negative change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 12 and 24
Population: Intent to treat (ITT) population included all participants randomized to the treatment group assigned, regardless of starting treatment or changing treatment during the study. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
unit on a scale
  Baseline: number analyzed (Participants) | 19 | 24
  Baseline | 1.22 (0.661) | 1.04 (0.595)
  Change from Baseline to Week 12: number analyzed (Participants) | 15 | 22
  Change from Baseline to Week 12 | -0.02 (0.348) | 0.24 (0.656)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 23
  Change from Baseline to Week 24 | 0.03 (0.449) | 0.41 (0.674)
Statistical Analysis 1: Comparison: Cenicriviroc 150 mg vs Placebo; Change from Baseline to Week 12; Test type: Other — This was a proof of concept study, and is not powered for statistical detection of differences between groups, no adjustments for multiplicity was made, or no-imputation for missing data; p = 0.2483, ANCOVA — An analysis of covariance (ANCOVA) model that included treatment and presence or absence of nonalcoholic steatohepatitis (NASH) as factors, and the baseline value of Matsuda index as a covariate was used for analysis; LS Mean Difference = -0.2286, 95% CI 2-sided [-0.62 to 0.17], Standard Error of Mean 0.195
Statistical Analysis 2: Comparison: Cenicriviroc 150 mg vs Placebo; Change form Baseline to Week 24; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.053, ANCOVA — An ANCOVA model that included treatment and presence or absence of NASH as factors, and the baseline value of Matsuda index as a covariate was used for analysis; LS Mean Difference = -0.4113, 95% CI 2-sided [-0.83 to 0.01], Standard Error of Mean 0.205

2. Primary Outcome: Change From Baseline in Adipose Tissue Insulin Resistance (Adipo-IR ) Index
Description: Change in adipose insulin sensitivity was measured by Adipo-IR. Adipo-IR= (Fasting Serum free fatty acid (FFA) mmol/L x FPI μIU/mL). A higher Adipo-IR index indicates the worst disease state. A lower Adipo-IR Index is best. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 12 and 24
Population: ITT population included all participants randomized to the treatment group assigned, regardless of starting treatment or changing treatment during the study. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
unit on a scale
  Baseline: number analyzed (Participants) | 18 | 23
  Baseline | 17.77 (14.074) | 17.74 (9.406)
  Change from Baseline to Week 12: number analyzed (Participants) | 14 | 22
  Change from Baseline to Week 12 | -1.41 (9.009) | -0.52 (8.745)
  Change from Baseline to Week 24: number analyzed (Participants) | 14 | 22
  Change from Baseline to Week 24 | -0.29 (7.524) | -4.22 (11.612)
Statistical Analysis 1: Comparison: Cenicriviroc 150 mg vs Placebo; Change from Baseline to Week 12; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.5297, ANCOVA — An ANCOVA model that included treatment and presence or absence of NASH as factors, and the baseline value of ADIPO-IR as a covariate was used for analysis; LS Mean Difference = -1.505, 95% CI 2-sided [-6.33 to 3.32], Standard Error of Mean 2.369
Statistical Analysis 2: Comparison: Cenicriviroc 150 mg vs Placebo; Change from Baseline to Week 24; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.2522, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS Mean Difference = 3.2146, 95% CI 2-sided [-2.4 to 8.83], Standard Error of Mean 2.757

3. Secondary Outcome: Change From Baseline in Macrophage Infiltration in Subcutaneous Adipose Tissue
Description: Macrophage infiltration in adipose tissue was assessed in paraffin-embedded adipose punch biopsies by immunohistochemistry stained for cluster of differentiation 68 (CD68), cluster of differentiation 163 (CD163), C-C chemokine receptor type 2 (CCR2), C-C chemokine receptor type 5 (CCR5) and cluster of differentiation 206 (CD206). A reduction in infiltration indicates less inflammation. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Week 24
Population: Safety Population included all participants who received at least one dose of study drug. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Median (Inter-Quartile Range); unit: cells/μL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 16 | 24
cells/μL
  CD68+, Baseline | 4.0 [2.0 to 5.0] | 3.0 [1.5 to 4.0]
  CD68+, Change from BL to Week 24 | 1.0 [-1.5 to 3.0] | 1.0 [-0.5 to 1.5]
  CD163+, Baseline | 9.5 [7.5 to 11.5] | 10.5 [7.0 to 19.0]
  CD163+, Change from BL at Week 24 | 2.0 [-1.0 to 6.5] | 1.0 [-3.5 to 4.0]
  CCR2+, Baseline | 10.0 [6.0 to 13.5] | 10.5 [7.0 to 17.0]
  CCR2+, Change from BL to Week 24 | 0.0 [-2.5 to 8.0] | 2.0 [-3.5 to 6.0]
  CCR5+, Baseline | 3.0 [2.0 to 4.0] | 3.0 [1.5 to 5.0]
  CCR5+, Change from BL to Week 24 | 1.0 [-1.0 to 2.0] | 0.0 [-1.5 to 1.5]
  CD206+, Baseline | 6.0 [4.0 to 10.5] | 7.0 [5.0 to 9.0]
  CD206+, Change from BL to Week 24 | 0.0 [-3.5 to 2.0] | -0.5 [-2.5 to 2.5]

4. Secondary Outcome: Change From Baseline in C-C Chemokine Receptor Type 2 (CCR2) and C-C Chemokine Receptor Type 5 (CCR5) in Subcutaneous Adipose Tissue
Description: CCR2 and CCR5 corresponding ligands' messenger ribonucleic acid (mRNA) gene expression were assessed in frozen adipose tissue by quantitative polymerase chain reaction (PCR). A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Week 24
Population: Safety Population included all participants who received at least one dose of study drug. Number analyzed is the number of participants with data available at the given timepoint
Measure: Median (Inter-Quartile Range); unit: copies per sample
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 15 | 21
copies per sample
  CCR2, Baseline: number analyzed (Participants) | 10 | 17
  CCR2, Baseline | 13.0 [6.75 to 16.5] | 13.7 [4.37 to 16.9]
  CCR2, Change from Baseline to Week 24: number analyzed (Participants) | 10 | 17
  CCR2, Change from Baseline to Week 24 | 2.6 [0.5 to 4.6] | 0.8 [-2.7 to 1.8]
  CCR5, Baseline: number analyzed (Participants) | 11 | 17
  CCR5, Baseline | 12.7 [8.19 to 17.3] | 15.2 [4.75 to 17.8]
  CCR5, Change from Baseline to Week 24: number analyzed (Participants) | 11 | 17
  CCR5, Change from Baseline to Week 24 | 3.6 [-0.7 to 5.2] | 0.1 [-1.6 to 1.0]

5. Secondary Outcome: Change From Baseline in Peripheral Monocyte Subsets (CD14/CD16)
Description: Peripheral monocyte subsets (cluster of differentiation 14 (CD14/cluster of differentiation 16 (CD16)] were measured in fresh peripheral blood mononuclear cells (PBMCs) samples by flow cytometry. Monocyte results are reported for Total, Classical (CD14+CD16-), Intermediate (CD14+CD16+) and Non-classical (CD14lowCD16+). A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: cells/μL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 15 | 21
cells/μL
  Total Monocytes, Baseline (BL) | 400 [200 to 400] | 400 [400 to 500]
  Total Monocytes, Change from Baseline to Week 24 | 0 [-200 to 0] | 0 [-100 to 0]
  Classical Monocytes, Baseline | 258 [179 to 368] | 351 [321 to 468]
  Classical Monocytes, Change from BL to Week 24 | -43.6 [-132 to 14.2] | -31 [-91 to 18]
  Intermediate Monocytes, Baseline | 16.8 [14.6 to 23.6] | 22.4 [11.8 to 32.0]
  Intermediate Monocytes, Change from BL to Week 24 | -1.4 [-10.2 to 2.5] | 3.8 [-4.7 to 25.8]
  Non-Classical Monocytes, Baseline | 24.9 [16.8 to 42.3] | 30.9 [18.4 to 46.1]
  Non-Classical Monocytes, Change from BL to Week 24 | -7.1 [-15.4 to 0] | -2.4 [-16.6 to 1.7]

6. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: A fasting blood sample was collected and was sent to a central laboratory for analysis of glucose. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day1) to Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
mg/dL
  Baseline | 119.55 (28.849) | 122.84 (33.212)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 24
  Change from Baseline to Week 12 | -5.56 (24.328) | -3.96 (24.412)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 24
  Change from Baseline to Week 24 | -3.25 (19.206) | -7.83 (25.610)

7. Secondary Outcome: Change From Baseline in Fasting Plasma Insulin (FPI)
Description: A fasting blood sample was collected and was sent to a central laboratory for analysis of insulin. A positive change from Baseline indicates improvement and a negative change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μIU/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
μIU/mL
  Baseline: number analyzed (Participants) | 19 | 24
  Baseline | 33.42 (26.427) | 33.38 (24.135)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 12 | -1.56 (10.204) | -5.26 (19.412)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 23
  Change from Baseline to Week 24 | -0.27 (8.464) | -6.83 (18.312)

8. Secondary Outcome: Change From Baseline in Quantitative Insulin Sensitivity Check Index (QUICKI)
Description: QUICKI is used to measure insulin sensitivity. QUICKI = 1/(log FPI μIU/mL + log FPG mg/dL). A positive change from Baseline indicates improvement and a negative change from Baseline indicates a worsening.
Time Frame: Baseline (Day1) to Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
unit on a scale
  Baseline: number analyzed (Participants) | 19 | 24
  Baseline | 0.29 (0.025) | 0.29 (0.023)
  Change from Baseline to Week 12: number analyzed (Participants) | 14 | 23
  Change from Baseline to Week 12 | 0.00 (0.018) | 0.00 (0.020)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 23
  Change from Baseline to Week 24 | 0.01 (0.019) | 0.01 (0.020)

9. Secondary Outcome: Change From Baseline in Homeostasis Model of Insulin Resistance (HOMA-IR)
Description: HOMA-IR = (FPG mg/dL x FPI μIU/mL)/405. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
unit on a scale
  Baseline: number analyzed (Participants) | 19 | 24
  Baseline | 10.56 (10.407) | 10.29 (8.931)
  Change from Baseline to Week 12: number analyzed (Participants) | 14 | 23
  Change from Baseline to Week 12 | -0.49 (3.182) | -1.96 (8.513)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 23
  Change from Baseline to Week 24 | -0.11 (3.170) | -3.07 (7.222)

10. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment of β-cell Function (HOMA-%B)
Description: HOMA-%B= (20 × FPI)/(FPG - 3.5). A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
unit on a scale
  Baseline: number analyzed (Participants) | 19 | 24
  Baseline | 5.63 (3.577) | 5.77 (4.079)
  Change from Baseline to Week 12: number analyzed (Participants) | 15 | 23
  Change from Baseline to Week 12 | -0.02 (1.795) | -0.74 (2.649)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 23
  Change from Baseline to Week 24 | -0.15 (1.304) | -0.73 (3.036)

11. Secondary Outcome: Change From Baseline in Fasting Glycosylated Hemoglobin A1c (HbA1c)
Description: as for outcome 6
Time Frame: Baseline (Day 1) to Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of HbA1c
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
percentage of HbA1c
  Baseline | 6.09 (0.735) | 6.23 (0.778)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 24
  Change from Baseline to Week 12 | -0.12 (0.634) | 0.09 (0.379)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 24
  Change from Baseline to Week 24 | -0.11 (0.567) | 0.00 (0.503)

12. Secondary Outcome: Change From Baseline in Plasma Glucagon Concentration
Description: A fasting blood sample was collected and was sent to a central laboratory for analysis of glucagon. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
ng/mL
  Baseline: number analyzed (Participants) | 19 | 24
  Baseline | 154.26 (32.877) | 169.13 (36.591)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 12 | 20.25 (23.251) | 4.61 (36.505)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 21
  Change from Baseline to Week 24 | 19.07 (35.977) | 19.14 (53.373)

13. Secondary Outcome: Plasma Glucose at 30, 60, 90 and 120 Minutes Following Glucose Load
Description: Blood was collected during the oral glucose tolerance test and was sent to a central laboratory for analysis of glucose.
Time Frame: Prior to Glucose Load, 30, 60, 90 and 120 minutes after glucose load on Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
mg/dL
  Week 12: Prior to Glucose Load: number analyzed (Participants) | 16 | 23
  Week 12: Prior to Glucose Load | 107.88 (12.638) | 119.39 (28.800)
  Week 12: 30 minutes: number analyzed (Participants) | 15 | 21
  Week 12: 30 minutes | 193.93 (32.458) | 205.90 (50.327)
  Week 12: 60 minutes: number analyzed (Participants) | 16 | 23
  Week 12: 60 minutes | 201.44 (49.884) | 232.74 (62.174)
  Week 12: 90 minutes: number analyzed (Participants) | 16 | 23
  Week 12: 90 minutes | 173.56 (56.169) | 227.00 (76.041)
  Week 12: 120 minutes: number analyzed (Participants) | 16 | 23
  Week 12: 120 minutes | 158.38 (46.411) | 201.04 (82.832)
  Week 24: Prior to Glucose Load: number analyzed (Participants) | 15 | 24
  Week 24: Prior to Glucose Load | 111.47 (20.035) | 114.88 (39.591)
  Week 24: 30 minutes: number analyzed (Participants) | 15 | 23
  Week 24: 30 minutes | 198.60 (44.223) | 198.65 (59.787)
  Week 24: 60 minutes: number analyzed (Participants) | 15 | 23
  Week 24: 60 minutes | 214.93 (58.414) | 232.09 (66.036)
  Week 24: 90 minutes: number analyzed (Participants) | 15 | 23
  Week 24: 90 minutes | 187.20 (53.835) | 220.61 (78.385)
  Week 24: 120 minutes: number analyzed (Participants) | 15 | 23
  Week 24: 120 minutes | 165.73 (53.378) | 191.26 (86.539)

14. Secondary Outcome: Plasma Insulin at 30, 60, 90 and 120 Minutes Following Glucose Load
Description: Blood was collected during the oral glucose tolerance test and was sent to a central laboratory for analysis of insulin.
Time Frame: Pre-glucose load, 30, 60, 90 and 120 minutes after glucose load on Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μIU/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
μIU/mL
  Week 12: Prior to Glucose Load: number analyzed (Participants) | 17 | 24
  Week 12: Prior to Glucose Load | 25.94 (12.065) | 27.96 (14.366)
  Week 12: 30 minutes: number analyzed (Participants) | 17 | 23
  Week 12: 30 minutes | 168.71 (61.276) | 170.83 (162.459)
  Week 12: 60 minutes: number analyzed (Participants) | 17 | 24
  Week 12: 60 minutes | 211.76 (72.218) | 203.29 (168.986)
  Week 12: 90 minutes: number analyzed (Participants) | 17 | 24
  Week 12: 90 minutes | 204.47 (108.028) | 236.63 (168.861)
  Week 12: 120 minutes: number analyzed (Participants) | 17 | 24
  Week 12: 120 minutes | 218.71 (158.013) | 223.96 (172.155)
  Week 24: Prior to Glucose Load: number analyzed (Participants) | 16 | 24
  Week 24: Prior to Glucose Load | 25.25 (15.571) | 26.54 (12.608)
  Week 24: 30 minutes: number analyzed (Participants) | 16 | 23
  Week 24: 30 minutes | 172.31 (78.152) | 145.26 (106.082)
  Week 24: 60 minutes: number analyzed (Participants) | 16 | 23
  Week 24: 60 minutes | 219.63 (134.629) | 217.57 (181.115)
  Week 24: 90 minutes: number analyzed (Participants) | 16 | 23
  Week 24: 90 minutes | 218.06 (105.188) | 233.22 (175.669)
  Week 24: 120 minutes: number analyzed (Participants) | 16 | 23
  Week 24: 120 minutes | 216.00 (119.872) | 265.00 (287.361)

15. Secondary Outcome: Change From Baseline in Area Under the Concentration-time Curve From Time 0 to 120 Minutes [AUC (0-120 Min)] for Serum Glucose
Description: AUC(0-120 min) was derived from the serum glucose values obtained during the oral glucose tolerance test. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Pre-glucose load) to 30, 60, 90 and 120 minutes after glucose load on Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes (min)*mg/dL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
minutes (min)*mg/dL
  Baseline: number analyzed (Participants) | 20 | 23
  Baseline | 22601 (6423) | 24977 (5543)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 21
  Change from Baseline to Week 12 | -1071 (4098) | -1031 (3322)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 21
  Change from Baseline to Week 24 | 329 (4883) | -1085 (4178)

16. Secondary Outcome: Change From Baseline in Area Under the Concentration-time Curve From Time 30 to 120 Minutes [AUC (30-120 Min)] for Serum Glucose
Description: AUC(30-120 min) was derived from the serum glucose values obtained during the oral glucose tolerance test. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Pre-glucose load) to 30, 60, 90 and 120 minutes after glucose load on Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes (min)*mg/dL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
minutes (min)*mg/dL
  Baseline: number analyzed (Participants) | 20 | 23
  Baseline | 17816 (5488) | 20097 (4620)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 20
  Change from Baseline to Week 12 | -941 (3490) | -923 (3092)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 21
  Change from Baseline to Week 24 | 383 (4380) | -889 (3497)

17. Secondary Outcome: Change From Baseline in AUC (0-120 Min) for Plasma Insulin
Description: AUC(0-120 min) was derived from the plasma insulin values obtained during the oral glucose tolerance test. A positive change from Baseline indicates improvement and a negative change from Baseline indicates a worsening.
Time Frame: Baseline (Pre-glucose load) to 30, 60, 90 and 120 minutes after glucose load on Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min*μIU/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
min*μIU/mL
  Baseline: number analyzed (Participants) | 19 | 24
  Baseline | 21261 (10716) | 24411 (13942)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 12 | 640 (6340) | -1850 (6916)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 22
  Change from Baseline to Week 24 | 2101 (8088) | -1703 (9109)

18. Secondary Outcome: Change From Baseline in AUC (30-120 Min) for Plasma Insulin
Description: AUC(30-120 min) was derived from the plasma insulin values obtained during the oral glucose tolerance test. A positive change from Baseline indicates improvement and a negative change from Baseline indicates a worsening.
Time Frame: Baseline (Pre-glucose load) to 30, 60, 90 and 120 minutes after glucose load on Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min*μIU/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
min*μIU/mL
  Baseline: number analyzed (Participants) | 19 | 24
  Baseline | 18178 (9082) | 21583 (12626)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 22
  Change from Baseline to Week 12 | 472 (5730) | -1830 (6532)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 22
  Change from Baseline to Week 24 | 1818 (7506) | -1467 (8523)

19. Secondary Outcome: Change From Baseline in Fasting Free Fatty Acids
Description: A fasting blood sample was collected and was sent to a central laboratory for analysis of free fatty acids. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
mg/dL
  Baseline: number analyzed (Participants) | 19 | 24
  Baseline | 15.36 (5.708) | 17.41 (6.913)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 12 | -0.74 (5.214) | 0.31 (7.489)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 23
  Change from Baseline to Week 24 | -0.09 (6.466) | -2.65 (8.856)

20. Secondary Outcome: Change From Baseline in Serum Adiponectin Concentration
Description: A fasting blood sample was collected and was sent to a central laboratory for analysis of adiponectin. A positive change from Baseline indicates improvement and a negative change from Baseline indicates a worsening.
Time Frame: Baseline (Day1) to Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
μg/mL
  Baseline: number analyzed (Participants) | 20 | 24
  Baseline | 3.99 (2.162) | 4.50 (2.253)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 23
  Change from Baseline to Week 12 | -0.01 (0.465) | 0.01 (0.937)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 24 | 0.64 (2.693) | -0.82 (2.222)

21. Secondary Outcome: Change From Baseline in Serum Resistin Concentration
Description: A fasting blood sample was collected and was sent to a central laboratory for analysis of resistin. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
ng/mL
  Baseline: number analyzed (Participants) | 20 | 24
  Baseline | 10.46 (3.724) | 10.44 (4.422)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 23
  Change from Baseline to Week 12 | -0.49 (3.019) | 0.10 (3.316)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 24 | -0.01 (4.168) | -1.19 (2.957)

22. Secondary Outcome: Serum FFA at 30, 60, 90 and 120 Minutes Following Glucose Load
Description: Blood was collected during the oral glucose tolerance test and was sent to a central laboratory for analysis of FFA.
Time Frame: Pre-glucose load, 30, 60, 90 and 120 minutes after glucose load on Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
mg/dL
  Week 12: Prior to Glucose Load: number analyzed (Participants) | 16 | 24
  Week 12: Prior to Glucose Load | 15.60 (5.578) | 17.44 (5.620)
  Week 12: 30 minutes: number analyzed (Participants) | 17 | 23
  Week 12: 30 minutes | 12.01 (5.464) | 14.24 (3.783)
  Week 12: 60 minutes: number analyzed (Participants) | 17 | 24
  Week 12: 60 minutes | 6.63 (3.925) | 8.85 (2.702)
  Week 12: 90 minutes: number analyzed (Participants) | 17 | 24
  Week 12: 90 minutes | 4.16 (3.104) | 5.43 (2.424)
  Week 12: 120 minutes: number analyzed (Participants) | 17 | 24
  Week 12: 120 minutes | 2.52 (1.378) | 4.08 (2.057)
  Week 24: Prior to Glucose Load: number analyzed (Participants) | 16 | 24
  Week 24: Prior to Glucose Load | 16.62 (4.162) | 14.60 (5.089)
  Week 24: 30 minutes: number analyzed (Participants) | 16 | 23
  Week 24: 30 minutes | 13.05 (5.059) | 12.84 (3.590)
  Week 24: 60 minutes: number analyzed (Participants) | 16 | 23
  Week 24: 60 minutes | 7.41 (3.462) | 8.23 (3.376)
  Week 24: 90 minutes: number analyzed (Participants) | 16 | 23
  Week 24: 90 minutes | 4.17 (2.238) | 5.66 (2.545)
  Week 24: 120 minutes: number analyzed (Participants) | 16 | 23
  Week 24: 120 minutes | 2.73 (1.092) | 4.05 (2.749)

23. Secondary Outcome: Change From Baseline in AUC (0-120 Min) for Serum FFA
Description: AUC(0-120 min) was derived from the serum FFA values obtained during the oral glucose tolerance test. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Pre-glucose load) to 30, 60, 90 and 120 minutes after glucose load on Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min*mmol/L
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
min*mmol/L
  Baseline: number analyzed (Participants) | 19 | 23
  Baseline | 37.2 (14.27) | 42.9 (14.57)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 22
  Change from Baseline to Week 12 | -5.4 (10.16) | -1.3 (14.46)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 21
  Change from Baseline to Week 24 | -3.4 (11.74) | -4.2 (18.98)

24. Secondary Outcome: Change From Baseline in AUC (30-120 Min) for Serum FFA
Description: AUC(30-120 min) was derived from the serum FFA values obtained during the oral glucose tolerance test. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Pre-glucose load) to 30, 60, 90 and 120 minutes after glucose load on Weeks 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min*mmol/L
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
min*mmol/L
  Baseline: number analyzed (Participants) | 20 | 23
  Baseline | 23.3 (11.55) | 25.6 (8.59)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 21
  Change from Baseline to Week 12 | -5.0 (7.49) | -0.9 (8.65)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 21
  Change from Baseline to Week 24 | -4.2 (8.61) | -1.5 (11.08)

25. Secondary Outcome: Change From Baseline in the Nonalcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS)
Description: Liver biopsy were performed during Screening and at Week 24 only for participants diagnosed with NASH. NAFLD activity score was determined based on 3 components: steatosis (0=<5% to 3=>66%), lobular inflammation (0=no foci to 3=>4 foci/200x) and hepatocellular ballooning (0=none to 2= many cells/prominent ballooning) for a total possible score of 0 to 8. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Screening) to Week 24
Population: ITT population included all participants randomized to the treatment group assigned, regardless of starting treatment or changing treatment during the study. Only participants confirmed at Screening with NASH by biopsy and had a biopsy conducted at Week 24 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 6 | 12
score on a scale
  Baseline | 4.33 (0.816) | 4.00 (1.279)
  Change from Baseline to Week 24 | -1.00 (1.265) | -0.33 (1.670)

26. Secondary Outcome: Number of Participants by NASH Clinical Research Network (CRN) Staging Categories
Description: Liver biopsy were performed during Screening and at Week 24 for participants diagnosed with NASH. The NASH CRN Brunt/Kleiner Fibrosis Staging System Fibrosis Stages are: 0 (None), 1 (Perisinusoidal or periportal), 1A (Mild, zone 3, perisinusoidal), 1B (Moderate, zone 3, perisinusoidal), 1C (Portal/periportal), 2 (Perisinusoidal and portal/periportal), 3 (Bridging fibrosis) and 4 (Cirrhosis).
Time Frame: Baseline (Screening) and Week 24
Population: ITT population included all participants randomized to the treatment group assigned, regardless of starting treatment or changing treatment during the study. Only participants confirmed at Screening with NASH by biopsy and had a biopsy conducted at Week 24 were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 6 | 12
Participants
  Baseline: Stage 0 | 2 | 0
  Baseline: Stage 1 | 2 | 7
  Baseline: Stage 1A | 1 | 3
  Baseline: Stage 1B | 0 | 0
  Baseline: Stage 1C | 0 | 0
  Baseline: Stage 2 | 0 | 2
  Baseline: Stage 3 | 1 | 0
  Baseline: Stage 4 | 0 | 0
  Week 24: Stage 0 | 2 | 4
  Week 24: Stage 1 | 3 | 6
  Week 24: Stage 1A | 0 | 2
  Week 24: Stage 1B | 0 | 0
  Week 24: Stage 1C | 0 | 0
  Week 24: Stage 2 | 0 | 0
  Week 24: Stage 3 | 1 | 0
  Week 24 : Stage 4 | 0 | 0

27. Secondary Outcome: Change From Baseline in Serum C-C Chemokine Receptor Type 2 (CCR2) Ligand: Monocyte Chemotactic Protein 1 (MCP-1)
Description: Blood was collected and was sent to a central laboratory for analysis of MCP-1. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 2, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
pg/mL
  Baseline: number analyzed (Participants) | 20 | 24
  Baseline | 445.86 (140.656) | 408.19 (117.099)
  Change from Baseline to Week 2: number analyzed (Participants) | 19 | 23
  Change from Baseline to Week 2 | 1333.68 (497.505) | 37.58 (71.741)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 23
  Change from Baseline to Week 12 | 1461.98 (663.465) | 31.98 (80.034)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 24 | 1248.86 (661.883) | 13.87 (79.726)

28. Secondary Outcome: Change From Baseline in Serum C-C Chemokine Receptor Type 5 (CCR5) Ligand: RANTES
Description: Blood was collected and was sent to a central laboratory for analysis of RANTES (regulated on activation normal T-cell expressed and secreted). A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 2, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
ng/mL
  Baseline: number analyzed (Participants) | 20 | 24
  Baseline | 36.95 (19.267) | 46.33 (28.419)
  Change from Baseline to Week 2: number analyzed (Participants) | 19 | 23
  Change from Baseline to Week 2 | -1.53 (20.643) | -1.13 (20.726)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 23
  Change from Baseline to Week 12 | -2.53 (18.729) | 0.65 (19.310)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 24 | -2.13 (29.003) | -5.35 (28.724)

29. Secondary Outcome: Change From Baseline in Serum CCR5 Ligand: Macrophage Inflammatory Protein 1 Alpha (MIP-1α)
Description: Blood was collected and was sent to a central laboratory for analysis of MIP-1α. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 2, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
pg/mL
  Baseline: number analyzed (Participants) | 20 | 24
  Baseline | 69.66 (20.275) | 62.85 (15.737)
  Change from Baseline to Week 2: number analyzed (Participants) | 19 | 23
  Change from Baseline to Week 2 | 64.11 (21.811) | -0.11 (8.583)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 23
  Change from Baseline to Week 12 | 63.75 (21.811) | -6.28 (10.135)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 24 | 61.08 (18.224) | -2.79 (9.445)

30. Secondary Outcome: Change From Baseline in Serum CCR5 Ligand: Macrophage Inflammatory Protein 1 Beta (MIP-1β)
Description: Blood was collected and was sent to a central laboratory for analysis of MIP-1β. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 2, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
pg/mL
  Baseline: number analyzed (Participants) | 20 | 24
  Baseline | 120.59 (40.483) | 102.85 (41.424)
  Change from Baseline to Week 2: number analyzed (Participants) | 19 | 23
  Change from Baseline to Week 2 | 163.26 (77.537) | 1.06 (15.232)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 23
  Change from Baseline to Week 12 | 152.21 (67.341) | -3.04 (20.482)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 24 | 147.83 (58.465) | -7.42 (15.499)

31. Secondary Outcome: Change From Baseline in Biomarker of Inflammation: Interleukin 1 Beta (IL-1β)
Description: Blood was collected and was sent to a central laboratory for analysis of IL-1β. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 2, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
pg/mL
  Baseline: number analyzed (Participants) | 20 | 24
  Baseline | 0.08 (0.058) | 0.20 (0.413)
  Change from Baseline to Week 2: number analyzed (Participants) | 19 | 23
  Change from Baseline to Week 2 | -0.03 (0.082) | -0.16 (0.413)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 23
  Change from Baseline to Week 12 | -0.01 (0.100) | -0.17 (0.418)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 24 | -0.03 (0.071) | -0.14 (0.420)

32. Secondary Outcome: Change From Baseline in Biomarker of Inflammation: Interleukin 6 (IL-6)
Description: Blood was collected and was sent to a central laboratory for analysis of IL-6. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 2, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
pg/mL
  Baseline: number analyzed (Participants) | 20 | 24
  Baseline | 3.54 (3.208) | 3.68 (2.274)
  Change from Baseline to Week 2: number analyzed (Participants) | 19 | 23
  Change from Baseline to Week 2 | -0.67 (2.885) | -0.11 (2.091)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 23
  Change from Baseline to Week 12 | -0.88 (3.299) | 0.20 (3.018)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 24 | -1.18 (2.958) | 1.08 (6.017)

33. Secondary Outcome: Change From Baseline in Biomarker of Inflammation: Interleukin 8 (IL-8)
Description: Blood was collected and was sent to a central laboratory for analysis of IL-8. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 2, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
pg/mL
  Baseline: number analyzed (Participants) | 20 | 24
  Baseline | 21.99 (8.454) | 18.42 (5.669)
  Change from Baseline to Week 2: number analyzed (Participants) | 19 | 23
  Change from Baseline to Week 2 | 0.55 (7.982) | 3.29 (7.846)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 23
  Change from Baseline to Week 12 | 4.16 (9.739) | 0.44 (7.475)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 24 | 1.31 (6.228) | -0.45 (6.452)

34. Secondary Outcome: Change From Baseline in Biomarker of Inflammation: Interleukin 10 (IL-10)
Description: as for outcome 31
Time Frame: Baseline (Day 1) to Weeks 2, 12 and 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
pg/mL
  Baseline: number analyzed (Participants) | 20 | 24
  Baseline | 3.05 (0.908) | 3.06 (0.694)
  Change from Baseline to Week 2: number analyzed (Participants) | 19 | 23
  Change from Baseline to Week 2 | 0.20 (0.772) | 0.10 (0.861)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 23
  Change from Baseline to Week 12 | 0.07 (0.896) | -0.17 (0.979)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 24 | -0.61 (0.406) | -0.37 (0.897)

35. Secondary Outcome: Change From Baseline in Biomarker of Inflammation: High Sensitivity C Reactive Protein (Hs-CRP)
Description: Blood was collected and was sent to a central laboratory for analysis of hs-CRP. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 2, 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
mg/L
  Baseline: number analyzed (Participants) | 19 | 24
  Baseline | 6.39 (9.232) | 5.39 (7.421)
  Change from Baseline to Week 2: number analyzed (Participants) | 18 | 23
  Change from Baseline to Week 2 | -1.58 (4.642) | 0.12 (2.934)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 22
  Change from Baseline to Week 12 | -0.50 (8.402) | 2.33 (6.813)
  Change from Baseline to Week 24: number analyzed (Participants) | 15 | 23
  Change from Baseline to Week 24 | -1.35 (2.843) | 0.14 (5.615)

36. Secondary Outcome: Change From Baseline in Biomarker of Inflammation: Tumor Necrosis Factor Alpha (TNF-α)
Description: Blood was collected and was sent to a central laboratory for analysis of TNF-α. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Weeks 2, 12, 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
pg/mL
  Baseline: number analyzed (Participants) | 20 | 24
  Baseline | 12.78 (3.208) | 12.35 (2.526)
  Change from Baseline to Week 2: number analyzed (Participants) | 19 | 23
  Change from Baseline to Week 2 | 0.68 (2.577) | -0.43 (2.592)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 23
  Change from Baseline to Week 12 | 0.58 (2.894) | -0.69 (2.484)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 24 | -0.06 (2.320) | -0.97 (2.361)

37. Secondary Outcome: Change From Baseline in Noninvasive Metabolic Biomarker: Hyaluronic Acid
Description: Blood was collected and was sent to a central laboratory for analysis of Hyaluronic Acid. A positive change from Baseline indicates improvement and a negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
ng/mL
  Baseline: number analyzed (Participants) | 20 | 23
  Baseline | 24.65 (18.511) | 19.78 (7.740)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 22
  Change from Baseline to Week 24 | 12.69 (19.622) | 4.86 (15.743)

38. Secondary Outcome: Change From Baseline in Noninvasive Metabolic Biomarker: Cytokeratin-18 (CK-18) [M30 and M65]
Description: Blood was collected and was sent to a central laboratory for analysis of CK-18. A positive change from Baseline indicates improvement and a negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
U/L
  Baseline: number analyzed (Participants) | 20 | 23
  Baseline | 399.35 (352.261) | 485.72 (547.707)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 22
  Change from Baseline to Week 24 | 1.88 (235.362) | -88.00 (338.731)

39. Secondary Outcome: Change From Baseline in Noninvasive Metabolic Biomarker: Fibroblast Growth Factor-21 (FGF-21)
Description: Blood was collected and was sent to a central laboratory for analysis of FGF-21. A negative change from Baseline indicates improvement and a positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
pg/mL
  Baseline: number analyzed (Participants) | 20 | 23
  Baseline | 266.75 (119.590) | 406.91 (260.751)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 22
  Change from Baseline to Week 24 | -3.53 (156.894) | 427.38 (1925.089)

40. Secondary Outcome: Change From Baseline in Noninvasive Metabolic Biomarker: Mac-2 Binding Protein (Mac-2BP)
Description: Blood was collected and was sent to a central laboratory for analysis of Mac-2BP. A negative change from Baseline indicates improvement and a positive change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
ng/mL
  Baseline: number analyzed (Participants) | 20 | 23
  Baseline | 5440.50 (1829.772) | 7156.96 (5336.192)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 22
  Change from Baseline to Week 24 | 20.94 (967.192) | -844.77 (2231.155)

41. Secondary Outcome: Change From Baseline in Noninvasive Metabolic Serum Biomarker: Cluster of Differentiation (CD95)
Description: Blood was collected and was sent to a central laboratory for analysis of CD95. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
ng/mL
  Baseline: number analyzed (Participants) | 20 | 23
  Baseline | 10.99 (2.478) | 11.11 (1.737)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 22
  Change from Baseline to Week 24 | -0.34 (2.259) | -1.00 (2.085)

42. Secondary Outcome: Change From Baseline in Noninvasive Metabolic Marker: Alpha-fetoprotein (AFP)
Description: Blood was collected and was sent to a central laboratory for analysis of AFP. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline (Day 1) to Week 24
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
ng/mL
  Baseline: number analyzed (Participants) | 20 | 22
  Baseline | 3.10 (1.483) | 2.91 (1.925)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 21
  Change from Baseline to Week 24 | 0.00 (0.730) | -0.14 (0.727)

43. Secondary Outcome: Change From Baseline in Non-invasive Imaging by Multiparametric Magnetic Resonance Imaging (MRI) for Liver Disease (LiverMultiScan™) Test: Fat Fraction
Description: LiverMultiscan™ tests via MRI were obtained at Baseline and at Weeks 12 and 24. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline to Weeks 12 and 24
Population: ITT population included all participants randomized to the treatment group assigned, regardless of starting treatment or changing treatment during the study. LiverMultiScan™ tests were performed in a subset of participants at one site. Number analyzed were the participants with analysis values at specified time point.
Measure: Mean (Standard Deviation); unit: percentage of fat
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 7 | 10
percentage of fat
  Baseline | 15.21 (9.112) | 13.56 (7.987)
  Change from Baseline to Week 12: number analyzed (Participants) | 6 | 10
  Change from Baseline to Week 12 | -0.05 (1.822) | -2.75 (7.121)
  Change from Baseline to Week 24: number analyzed (Participants) | 5 | 10
  Change from Baseline to Week 24 | 1.08 (3.238) | -5.37 (7.486)

44. Secondary Outcome: Change From Baseline in Non-invasive Imaging by Multiparametric Magnetic Resonance Imaging (MRI) for Liver Disease (LiverMultiScan™) Test: Corrected T1 (cT1)
Description: LiverMultiscan™ via MRI were obtained at Baseline and at Weeks 12 and 24. The mean of 4 regions of interest as selected by the technician is reported. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline to Weeks 12 and 24
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: milliseconds (ms)
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 7 | 10
milliseconds (ms)
  Baseline | 923.72 (76.249) | 911.97 (88.007)
  Change from Baseline to Week 12: number analyzed (Participants) | 6 | 10
  Change from Baseline to Week 12 | -10.62 (22.211) | -5.60 (52.203)
  Change from Baseline to Week 24: number analyzed (Participants) | 5 | 10
  Change from Baseline to Week 24 | 0.03 (28.771) | -3.95 (55.402)

45. Secondary Outcome: Change From Baseline in Non-invasive Imaging by Multiparametric Magnetic Resonance Imaging (MRI) for Liver Disease (LiverMultiScan™) Test: cT1 Mode Values Within the Liver
Description: LiverMultiscan™ via MRI were obtained at Baseline and at Weeks 12 and 24. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline to Weeks 12 and 24
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 7 | 10
ms
  Baseline | 917.95 (68.147) | 901.67 (77.461)
  Change from Baseline to Week 12: number analyzed (Participants) | 6 | 10
  Change from Baseline to Week 12 | -15.37 (18.348) | -4.00 (42.298)
  Change from Baseline to Week 24: number analyzed (Participants) | 5 | 10
  Change from Baseline to Week 24 | -2.83 (18.707) | 0.89 (42.722)

46. Secondary Outcome: Change From Baseline in Non-invasive Imaging by Multiparametric Magnetic Resonance Imaging (MRI) for Liver Disease (LiverMultiScan™) Test: Liver Inflammation and Fibrosis (LIF) Score
Description: LiverMultiscan™ tests via MRI were obtained at Baseline and at Weeks 12 and 24. The mean of 4 regions of interest as selected by the technician is reported. The LIF Score ranges from 0=no liver disease to 4=severe liver disease. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline to Weeks 12 and 24
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 7 | 10
unit on a scale
  Baseline | 2.50 (0.853) | 2.34 (0.868)
  Change from Baseline to Week 12: number analyzed (Participants) | 6 | 10
  Change from Baseline to Week 12 | -0.11 (0.259) | -0.01 (0.450)
  Change from Baseline to Week 24: number analyzed (Participants) | 5 | 10
  Change from Baseline to Week 24 | 0.01 (0.345) | -0.00 (0.505)

47. Secondary Outcome: Change From Baseline in Non-invasive Imaging by Multiparametric Magnetic Resonance Imaging (MRI) for Liver Disease (LiverMultiScan™) Test: Iron Content
Description: LiverMultiscan™ tests via MRI were obtained at Baseline and at Weeks 12 and 24. A positive change from Baseline indicates improvement and a negative change from Baseline indicates a worsening.
Time Frame: Baseline to Weeks 12 and 24
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: mg/g of liver
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 7 | 10
mg/g of liver
  Baseline | 1.24 (0.151) | 1.29 (0.152)
  Change from Baseline to Week 12: number analyzed (Participants) | 6 | 10
  Change from Baseline to Week 12 | 0.03 (0.121) | -0.06 (0.117)
  Change from Baseline to Week 24: number analyzed (Participants) | 5 | 10
  Change from Baseline to Week 24 | 0.00 (0.122) | -0.14 (0.151)

48. Secondary Outcome: Change From Baseline in Body Weight
Description: A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline to Weeks 2, 4, 8, 12, 16, 20 and 24
Population: Safety Population included all participants who received at least one dose of study drug. Number analyzed were the participants with analysis values at specified time point.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
kg
  Baseline | 94.92 (14.282) | 100.92 (15.359)
  Change from Baseline to Week 2: number analyzed (Participants) | 19 | 23
  Change from Baseline to Week 2 | -0.22 (1.760) | -1.10 (2.008)
  Change from Baseline to Week 4: number analyzed (Participants) | 19 | 24
  Change from Baseline to Week 4 | -0.52 (2.417) | -1.43 (2.453)
  Change from Baseline to Week 8: number analyzed (Participants) | 18 | 24
  Change from Baseline to Week 8 | 0.21 (2.029) | -1.56 (3.162)
  Change from Baseline to Week 12: number analyzed (Participants) | 17 | 24
  Change from Baseline to Week 12 | 0.53 (2.967) | -1.50 (3.879)
  Change from Baseline to Week 16: number analyzed (Participants) | 16 | 24
  Change from Baseline to Week 16 | 0.87 (3.160) | -1.73 (4.018)
  Change from Baseline to Week 20: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 20 | 0.17 (3.555) | -2.15 (4.152)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 23
  Change from Baseline to Week 24 | 0.03 (3.656) | -2.44 (4.417)

49. Secondary Outcome: Change From Baseline in Liver Transaminase: Alanine Aminotransferase (ALT)
Description: Blood was collected and was sent to a central laboratory for analysis of ALT. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline to Weeks 12 and 24
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
U/L
  Baseline | 55.76 (42.044) | 51.28 (39.066)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 22
  Change from Baseline to Week 12 | -0.22 (14.621) | -6.88 (19.856)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 24
  Change from Baseline to Week 24 | 0.40 (21.223) | -8.95 (24.300)

50. Secondary Outcome: Change From Baseline in Liver Transaminase: Aspartate Aminotransferase (AST)
Description: Blood was collected and was sent to a central laboratory for analysis of AST. A negative change from Baseline indicates improvement and a positive change from Baseline indicates a worsening.
Time Frame: Baseline to Weeks 12 and 24
Population: as for outcome 48
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
U/L
  Baseline | 33.88 (17.885) | 36.10 (26.712)
  Change from Baseline to Week 12: number analyzed (Participants) | 16 | 22
  Change from Baseline to Week 12 | 0.46 (9.447) | -3.31 (16.374)
  Change from Baseline to Week 24: number analyzed (Participants) | 16 | 24
  Change from Baseline to Week 24 | 1.57 (13.022) | -3.75 (15.966)

51. Secondary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE)
Description: An AE is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is an AE that occurs or worsens after receiving study drug.
Time Frame: 24 weeks
Population: Safety Population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
Participants | 10 | 18

52. Secondary Outcome: Number of Participants With Clinically Relevant Changes From Baseline in Vital Signs
Description: Vital signs included Systolic Blood Pressure, Diastolic Blood Pressure, Heart Rate, Respiratory Rate and Temperature. The investigator determined if the vital sign measurements were clinically relevant.
Time Frame: 24 weeks
Population: Safety Population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
Participants | 0 | 0

53. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Electrocardiogram (ECG) Results
Description: A standard 12 lead ECG was performed. The investigator determined if the abnormal results were clinically significant.
Time Frame: Baseline 24 weeks
Population: Safety Population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
Participants | 0 | 0

54. Secondary Outcome: Plasma Cenicriviroc Concentrations
Time Frame: Baseline (Day 1) one sample predose; Weeks 2, 12 and 24 one sample predose and one sample postdose
Population: Pharmacokinetic (PK) Population included all participants in the safety population who received at least 1 dose of study drug and had at least 1 PK assessment.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cenicriviroc 150 mg
Number analyzed (Participants) | 20
ng/mL
  Baseline: Pre-Dose | 0.0 (0.00)
  Week 2: Pre-Dose: number analyzed (Participants) | 18
  Week 2: Pre-Dose | 168.7 (165.53)
  Week 2: Post-Dose: number analyzed (Participants) | 17
  Week 2: Post-Dose | 170.7 (182.87)
  Week 12: Pre-Dose: number analyzed (Participants) | 17
  Week 12: Pre-Dose | 383.3 (755.28)
  Week 12: Post-Dose: number analyzed (Participants) | 17
  Week 12: Post-Dose | 320.4 (623.34)
  Week 24: Pre-Dose: number analyzed (Participants) | 16
  Week 24: Pre-Dose | 230.7 (382.75)
  Week 24: Post-Dose: number analyzed (Participants) | 15
  Week 24: Post-Dose | 127.4 (92.26)

55. Secondary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: Physical examination included assessment of the following body systems: Abdomen, Cardiovascular, Extremities, Head, Eyes, Ears, Nose, Throat, Lungs, Lymph Nodes, Neurological, Skin and Thyroid. The number of participants with any abnormal findings at Baseline and participants with any abnormal findings Post-Baseline are reported.
Time Frame: 24 weeks
Population: Safety Population included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cenicriviroc 150 mg | Placebo
Number analyzed (Participants) | 20 | 25
Participants
  Baseline | 3 | 8
  Post-Baseline | 3 | 13

ADVERSE EVENTS:
Time Frame: First dose of study drug to within 28 days post last dose of study drug (Up to approximately 29 weeks)
Description: Safety Population included all participants who received at least one dose of study drug.
Arm/Group | Cenicriviroc 150 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/25
Other Adverse Events (participants affected / at risk) | 10/20 | 11/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cenicriviroc 150 mg (N=20) | Placebo (N=25)
Depression (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cenicriviroc 150 mg (N=20) | Placebo (N=25)
Constipation (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Bronchitis (Infections and infestations) | 1 | 0
Epididymitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
White blood cell count increased (Investigations) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Plantar fascial fibromatosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.